CLINICAL TRIAL: NCT04048590
Title: Skilled Nursing Facility Care at Home for Adults Discharged From the Hospital: A Pilot Randomized Controlled Evaluation
Brief Title: Skilled Nursing Facility at Home: A Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Spire Health, Inc. (Unknown); Reflexion Health, Inc. (Industry)
Responsible Party: Principal Investigator, David Levine, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019P001231
Record Dates: First submitted 2019-06-05; First posted 2019-08-07 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Skilled Nursing Facilities; Rehabilitation
Keywords: Skilled Nursing Facilities; Home-based care; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control subjects will receive care at a skilled nursing facility.
- Intervention (Active Comparator): Intervention subjects will go home from the hospital and receive care from a specialized care team.
  Interventions: Other: Skilled Nursing Facility at Home

INTERVENTIONS:
Other: Skilled Nursing Facility at Home — We plan to deploy an innovative and tailored set of rehabilitation services delivered in a patient's home that would allow for discharge from the hospital directly to home, despite the need for more intensive rehabilitative care not currently found in the home setting. We plan to combine a high-touch and high-tech approach that combines novel uses of personnel practicing at the very top of their license with novel uses of technology.
  Other Names: Rehab at Home
  Arms: Intervention

SUMMARY:
We seek to pilot a randomized controlled evaluation of skilled nursing facility care at home. We plan to enroll patients who would normally be sent to a skilled nursing facility following following hospitalization. As a substitute for a skilled nursing facility, we will deploy a technology-enabled team to the home to care for patients.

DETAILED DESCRIPTION:
Post-acute care (PAC) encompasses the wide range of rehabilitative services used to restore a patient's maximal functional status following discharge from an acute hospitalization with the goal of restoring healthful aging. Approximately 40% of all hospitalized Medicare beneficiaries utilize PAC, accounting for 20% of all Medicare expenditures. PAC is a fast-growing segment of Medicare, and for some conditions, Medicare spending on PAC nearly equals that of the initial hospitalization, with skilled nursing facility (SNF) PAC accounting for most of these trends. The quality of SNF PAC is suspect, with substantial regional variation, insufficient physical therapy delivery, high readmission rates, poor attention to whole-person care, and poor patient experience. Given these concerns, some experts have called for national improvement.

The investigators propose a home-based PAC model that substitutes for treatment in a traditional SNF PAC facility. We believe that rehabilitation following hospitalization in one's home has several benefits: support tailored to one's actual living circumstances, an environment that encourages earlier mobilization, support of and interaction with family and caregivers, and psychosocial benefits of being at home. To promote aging in place, the investigators plan to deploy an innovative and tailored set of SNF PAC services delivered in a patient's home that would allow for discharge from the hospital directly to home, despite the need for more intensive rehabilitative care not currently found in the home setting. The investigators plan to combine a high-touch and high-tech approach that combines novel uses of personnel practicing at the very top of their license (certified nursing assistants, nurses, home health aides) with novel uses of technology (virtual physical therapy with three-dimensional camera feedback, continuous monitoring, and video visits).

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* Requires skilled nursing facility care following hospitalization, as determined by inpatient team
* Lives within 10 miles of Brigham and Women's Hospital (BWH) or Brigham and Women's Faulkner Hospital (BWFH)
* Has capacity to consent
* Likely to return to community dwelling status
* Patient on medical service

  * Pending low volume, we reserve ability to phase in patients on surgical services, including orthopedic trauma

Exclusion Criteria:

* Social

  * Undomiciled
  * No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
  * In police custody
  * Resides in facility that does not allow advanced on-site medical care
  * Domestic violence screen positive
* Clinical

  * Requires care of new ostomy or teaching ostomy care associated with complication
  * Requires frequent suctioning, tracheostomy, and/or ventilator needs
  * Requires significant durable medical equipment not already in place at home (e.g., Hoyer lift)
  * Home unable to accommodate patient in current state as determined by the SNF-at-Home Checklist for Home
  * Acute delirium
  * End stage renal disease on hemodialysis
  * On methadone requiring daily pickup of medication
  * Requires administration of intravenous controlled substances
  * Requires administration of specialty medications not already in place at home
  * Requires transfusion of blood products
  * Requires multiple transfers back and forth to hospital for specialty medical care
* Home SNF census is full

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Cost of care | Enrollment to Discharge, up to 10 weeks
  Internal cost of providing rehabilitation care in dollars

SECONDARY OUTCOMES:
Length of stay | Enrollment to Discharge, up to 10 weeks
  Length of stay in days
Transfer back to the hospital | Enrollment to Discharge, up to 10 weeks
  Frequency of return to the hospital
Change in activities of daily living | Enrollment to Discharge, up to 10 weeks
  Change in activities of daily living from admission to discharge. Activities of daily living is a scale 0-6, with 6 representing more activities.
Change in instrumental activities of daily living | Enrollment to Discharge, up to 10 weeks
  Change in instrumental activities of daily living from admission to discharge. Instrumental activities of daily living is a scale 0-8, with 8 representing more activities.
Modified picker experience questionnaire | Discharge, up to 10 weeks
  Score on the modified picker experience questionnaire, with scores between 0-15, where 15 represents a higher/better score.
3 item care transition measure | Discharge, up to 10 weeks
  Score on the 3 item care transition measure, with scores between 0 and 12, where 12 represents a higher/better score.
Unplanned readmission rate | Enrollment to 30-days after discharge, up to 10 weeks
  Frequency of unplanned readmissions within 30-days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, MD, MPH, MA, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caplan GA, Coconis J, Board N, Sayers A, Woods J. Does home treatment affect delirium? A randomised controlled trial of rehabilitation of elderly and care at home or usual treatment (The REACH-OUT trial). Age Ageing. 2006 Jan;35(1):53-60. doi: 10.1093/ageing/afi206. Epub 2005 Oct 20. PMID 16239239
- [Background] David S, Sheikh F, Mahajan D, Greenough W, Bellantoni M. Whom Do We Serve? Describing the Target Population for Post-acute and Long-term Care, Focusing on Nursing Facility Settings, in the Era of Population Health in the United States. J Am Med Dir Assoc. 2016 Jul 1;17(7):574-80. doi: 10.1016/j.jamda.2016.05.004. No abstract available. PMID 27346649
- [Background] Mechanic R. Post-acute care--the next frontier for controlling Medicare spending. N Engl J Med. 2014 Feb 20;370(8):692-4. doi: 10.1056/NEJMp1315607. No abstract available. PMID 24552315
- [Background] Chandra A, Dalton MA, Holmes J. Large increases in spending on postacute care in Medicare point to the potential for cost savings in these settings. Health Aff (Millwood). 2013 May;32(5):864-72. doi: 10.1377/hlthaff.2012.1262. PMID 23650319
- [Derived] Levine DM, Cueva MA, Shi S, Limaj I, Wambolt B, Grabowski DC, Schnipper JL, Pu CT. Skilled Nursing Facility Care at Home for Adults Discharged From the Hospital: A Pilot Randomized Controlled Trial. J Appl Gerontol. 2022 Jun;41(6):1585-1594. doi: 10.1177/07334648221077092. Epub 2022 Mar 10. PMID 35266835